CLINICAL TRIAL: NCT04599179
Title: Stage IV Gastric Cancer: Patient's Quality of Life (QoL) After Surgical or Endoscopic Palliative Treatment.
Brief Title: SEMS and Gastroenterostomy
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, ENRICO FIORI, Professor of Surgery, University of Roma La Sapienza
Other Study IDs: 14102020
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients underwent placement of a self-expandable metal stent (SEMS)
  Interventions: Device: self-expandable metal stent
- Group 2: Patients underwent to stomach-partitioning gastrojejunostomy

INTERVENTIONS:
Device: self-expandable metal stent — self-expandable metal stent endoscopic positioning
  Other Names: stomach-partitioning gastrojejunostomy (SPGJ)
  Groups: Group 1

SUMMARY:
More than 20% of patients with gastric cancer have at presentation a stage IV disease. Advanced adenocarcinoma of the antro-pyloric region often determines a condition of gastric outlet obstruction syndrome (GOOS), which requires a rapid resolution for the severe consequences that will occur if the obstruction is not resolved. GOOS causes malnutrition, fluid and electrolyte imbalances that are difficult to control. Laparoscopic or open gastroenterostomy has been proposed as the treatment of choice in patients with advanced unresectable distal stomach tumor presenting with symptoms of GOOS. Noticeably, laparoscopic gastroenterostomy might be difficult to be performed in a hostile abdomen because of the involvement of the root of the mesentery, infiltration of the surrounding structures and peritoneal carcinosis. Furthermore, laparoscopic or open gastroenterostomy provides suboptimal palliation, because it is associated with postoperative complications ranging from 15% to 50% related to a delayed gastric emptying and a protract postoperative hospital stay. These results negatively affect the quality of life (QoL), and therefore, the efficacy of gastroenterostomy for palliation has been questioned. In 1997, Kaminishi et al. introduced a technique of stomach-partitioning gastrojejunostomy (SPGJ), which divides the lower part of the stomach and connects the jejunum to the proximal part of the stomach while maintaining a tunnel that is 2 to 3 cm in diameter along the lesser curvature. This technique theoretically provides some benefits: endoscopic evaluation of the tumor response to adjuvant chemotherapy and the possibility of repeated endoscopic local treatment on the tumor, prevention of ingested food retention in the distal part of the stomach thus facilitating gastric emptying and improving patient's QoL. A current alternative to laparoscopic or open surgical approach to an advanced gastric tumor is the positioning of a self-expandable metal stent (SEMS) which offers many potential advantages: the avoidance of general anaesthesia for a laparoscopic or open approach, a shorter hospital stay and a minor patient postoperative discomfort.

We want to perform a prospective longitudinal cohort trial, comparing the QoL of patients affected with stage IV antropyloric stomach cancer and symptoms of GOOS who underwent endoscopic placement of a SEMS or after open SPGJ.

ELIGIBILITY:
Inclusion criteria are age less than 85 years, pre-treatment histological diagnosis of gastric adenocarcinoma, computed tomographic (CT), adjuvant-neoadjuvant chemotherapy regimen, symptoms of GOOS (symptoms of GOOS include: regular, frequent feeling of bloating or fullness; feeling full after eating less food; nausea and vomiting of undigested food, especially right after eating, abdominal pain) lumen reduction ranging between 70% and 99% at gastroscopy.

Criteria for exclusion are a white blood cells count less than 4,000/L, a platelet count less than 70,000/L, patients with renal failure (i.e. albumin to creatinine ratio > 30 mg/mmol and estimated glomerular filtration rate < 30-44 mL/min/1.73m2), patients with major alterations of liver function tests (i.e. total bilirubin > 25.6 μmol/L, AST > 5 U/L, ALT >5 U/L, PT-INR > 1.5).

-

Ages: 30 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presenting with stage IV antropyloric gastric cancer at our Institution are enrolled
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL) after endoscopic or surgical treatment | 6-12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided